CLINICAL TRIAL: NCT02473081
Title: The Long-term Effect of a Minimal Psychological Intervention on Type 2 Diabetes Patients' Depressive Symptom, Diabetes-related Distress and Glycemic Control
Brief Title: Minimal Psychological Intervention in Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ching-Ju Chiu, Assistant Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NSC 101-2314-B-006-001-
Record Dates: First submitted 2015-06-09; First posted 2015-06-16 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2; Depression
Keywords: Type 2 diabetes; Minimal psychological intervention; Glycemic control; Depressive symptoms; Problem Area in Diabetes; Middle-aged and older adults; HbA1c protein, human
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Minimal Psychological Intervention (Experimental): Participants allocated to this group not only received the usual care as given by their family physicians, but also accepted biweekly minimal psychological intervention via telephone during six weeks.
  Interventions: Behavioral: Minimal psychological intervention; Other: Usual care
- Usual care (Other): Participants in this group received usual care only.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Minimal psychological intervention — Minimal psychological intervention (MPI) was used to help adults with chronic illness to manage their psychological burden by breaking through a negative spiral between thoughts and behaviors.
  Arms: Minimal Psychological Intervention
Other: Usual care — Usual care was given by their family physicians.

SUMMARY:
The purpose of this study is to determine whether the telephone-delivered Minimal Psychological Intervention (MPI) could improve diabetes' depressive symptom and diabetes-related immediately , as well as HbA1c level in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Diabetes disease

Exclusion Criteria:

* Were using anti-depression medication
* With ongoing psychological/psychiatric treatment
* Had been diagnosed with psychosis (ex. schizophrenia or bipolar disorder)
* Had severe cognitive problem or hearing impairment
* Lost their partner within three months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Depressive symptom assessed by CES-D 10 | At three points in time: at baseline (wave 1), post-intervention or 6 weeks after randomization (wave 2), and 1 month after the intervention period or 10 weeks after randomization (wave 3)
  Depressive symptom score was assessed with the 10-item Center for Epidemiologic Studies Depression Scale (CES-D 10).
Diabetes-related distress assessed by PAID scale | At three points in time: at baseline (wave 1), post-intervention or 6 weeks after randomization (wave 2), and 1 month after the intervention period or 10 weeks after randomization (wave 3)
  Diabetes-specific emotional distress was assessed with the Problem Areas in Diabetes (PAID) scale.
Hemoglobin A1c | Participants were measured during entire follow-up period, an average period of 3 months.